CLINICAL TRIAL: NCT06281951
Title: Nebulized Fentanyl in Healthy Volunteers : Comparison of Facial Versus Intranasal Aerosol Administration by Pharmacometric Modeling
Brief Title: Nebulized Fentanyl in Healthy Volunteers
Acronym: AEROfen
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2022/0271/HP
Record Dates: First submitted 2024-02-05; First posted 2024-02-28 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Analgesia; Emergencies
Keywords: Severe acute pain; Pharmacometry; Fentanyl; Emergency medicine; Pupillometry (PUAL); Non-invasive analgesia (Intranasal, Facial aerosol)
MeSH Terms: conditions — Agnosia; Emergencies; Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Facial Nebulization (Experimental): Fentanyl's facial nebulization in healthy volunteers.
  Interventions: Drug: Fentanyl - Inhalation by facial nebulization
- Intranasal (Experimental): Fentanyl's intranasal inhalation in healthy volunteers.
  Interventions: Drug: Fentanyl - Nebulisation

INTERVENTIONS:
Drug: Fentanyl - Inhalation by facial nebulization — 3 administrations based on a weight-dependent threshold (40 µg per administration for a weight < 70kg and 50 µg per administration for a weight ≥ 70kg).
  Other Names: AEROGEN Nebulizer
  Arms: Facial Nebulization
Drug: Fentanyl - Nebulisation — 3 administrations based on a weight-dependent threshold (20 µg/administration and for a weight < 70kg and 30 µg/administration for a weight ≥ 70kg). The dose of each bolus will be distributed at equivalent volume in both nasal pits
  Other Names: Teleflex intranasal device
  Arms: Intranasal

SUMMARY:
Pain constitutes the predominant motive prompting individuals to seek emergency medical attention, accounting for 80% of admissions to emergency departments. Presently, it is imperative to employ expeditious and efficacious analgesia-sedation methodologies, obviating the necessity for intravenous administration, while ensuring the secure delivery of pharmaceutical agents. The objective of this study is to assess the feasibility and comfort of nebulized intranasal or facial aerosol administration of Fentanyl through the implementation of a pharmacokinetic/pharmacodynamic (PK/PD) study

DETAILED DESCRIPTION:
The prompt identification, assessment, and management of pain are imperative in the context of emergency medicine, necessitating rapid and effective interventions. In the realm of pain management, the investigators deemed it crucial to concentrate on non-invasive approaches, such as opioid nebulization, while ensuring the safe and controlled delivery of the pharmaceutical agent. Intranasal analgesia emerges as a particularly suitable option due to its non-invasiveness, painlessness, ease of administration, cost-effectiveness, and lack of stringent aseptic requirements, making it especially convenient for patients in pain. However, the administration of medications in nasal drop form lacks precise control over the quantity of the active drug, potentially resulting in a hepatic first-pass effect and inactivation before systemic absorption, particularly with large quantities and subsequent swallowing.

Facial nebulization of opiates presents an alternative method for analgesic administration. Traditional pneumatic nebulizers, readily available in emergency settings, are economical aerosol generators. However, they pose challenges related to the reproducibility of administration and the potential for infectious contamination due to the dispersion of nebulized particles in the air between inhalations. Palladium vibrating screen aerosols, designed to produce optimal particle sizes for drug delivery to the lungs, show promise due to their more occlusive system, offering enhanced performance. Yet, these devices lack evaluation in the realm of opioids, particularly in terms of objective nociception measurement.

Pupillometry, specifically PUAL (pupillary unrest in ambient light), stands out as an objective technique capable of quantifying nociception or opioid impregnation. PUAL monitors variations in pupil diameter over time, and previous studies have indicated an inverse correlation between the analgesic response to opioid treatment and PUAL amplitude, suggesting it could serve as a marker of central opioid impregnation. However, scientific evidence in alert emergency medicine patients remains lacking. Additionally, standard clinical pharmacodynamic evaluation criteria for opioids are not well-suited to the variability of therapeutic responses in emergency situations.

Pharmacometric models offer a quantitative approach to understanding relationships between administered drugs, clinico-biological covariates, exposure, and responses (biomarkers, efficacy, safety) as they evolve over time in individual patients and populations. This pilot study aims to evaluate the feasibility, safety, effects, and robustness of nebulized fentanyl administration via facial aerosol or intranasal routes in a population of adult healthy volunteers, employing equivalent analgesic doses. PUAL will serve as an objective pharmacodynamic marker of central opioid impregnation, coupled with pharmacokinetic modeling of nebulized fentanyl administered via facial aerosol or intranasally. The development of a pharmacometric model using a population-based approach aims to establish fentanyl titration strategies based on the objective of reducing PUAL while ensuring central opioid impregnation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and < 68 years
* BMI between 19 and 29 kg/m²
* Affiliation to a social security scheme
* Adult who has read and understood the information letter and signed the consent form
* Woman capable of procreating (a woman is considered capable of procreating, i.e. fertile, after menarche and until she becomes menopausal, unless she is definitely sterile ) having very effective contraception (combined hormonal contraception (containing estrogens and progestins) associated with inhibition of ovulation, progestin-only hormonal contraception associated with inhibition of ovulation, intrauterine device, hormone-releasing intrauterine system (IUS), bilateral tubal occlusion, vasectomized partner, sexual abstinence) for 1 year and a negative urine pregnancy test at inclusion and during the duration of the study.
* Woman definitely surgically sterile (hysterectomy, bilateral salpingectomy and bilateral oophorectomy). Postmenopausal woman: The postmenopausal state is defined by the absence of periods for 12 months without any other medical cause.

Exclusion Criteria:

* Weight < 50 kg
* Taking long-term painkillers or narcotics
* Sharp pain
* Stable chronic pain (>3 months, with or without long-term treatment)
* Known chronic pathology stabilized or decompensated (hypertension, renal, cardiac, hepatic insufficiency, etc.)
* Stable or decompensated chronic respiratory pathology
* Chronic neuropsychiatric pathology likely to modify the pain threshold
* Long-term treatment with an action on the nervous system such as respiratory depression: benzodiazepines, neuroleptics, agonist/antagonist of the opioid system
* Treatment or toxicant whose association is not recommended with fentanyl (alcohol, cannabis, etc.)
* Central nervous system modulator treatment
* Pathologies blocking the pupillary response: Claude-Bernard-Horner syndrome, Adie syndrome, Argyll-Robertson pupil, senile miosis, dysautonomic neuropathy (advanced diabetes, systemic amyloidosis), cataract
* Treatment responsible for fluctuation in PUAL measurements: parasympathetic modulators (clonidine, dexmedetomidine, droperidol, metoclopramide)
* No-indication to FENTANYL PIRAMAL 100µg/2mL, solution for injection in ampoule
* No-indication to PROAMP SODIUM CHLORIDE 0.9%, solution for injection
* Ongoing treatment with nasal vasoconstrictors
* Peripheral oxygen saturation less than 93%
* Alteration of cognitive state: comprehension disorder, language disorder, memory disorder, confusion
* Deaf or mute patient
* Usual heart rate such as HR< 40 bpm and/or hypotension with systolic blood pressure SBP< 100 mm Hg
* Atrioventricular block on ECG
* History of cataract surgery
* Confirmed or suspected covid 19 / active flu infection less than 15 days old
* Allergy to plastic
* Pregnant or parturient or breastfeeding woman or proven absence of contraception
* Person deprived of liberty by an administrative or judicial decision or person placed under judicial protection/under guardianship or curatorship
* Person participating in research participating in another trial / having participated in another trial within 2 weeks
* History of illness or psychological or sensory abnormality likely to prevent the subject from fully understanding the conditions required for participation in the protocol or preventing them from giving informed consent

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of [F] bioavailability via facial nebulization and intranasal inhalation. | 6 hours
  Bioavailability [F] will be expressed as percent mean +/- standard deviation for each group.

SECONDARY OUTCOMES:
Measurement of maximum decrease in PUAL (pupillary under ambient light) between facial nebulization and intranasal inhalation. | 6 hours
  Maximum decrease in PUAL will be expressed as percent of baseline value +/- standard deviation for each group.
Measurement of the difference between observed and predicted PUAL values by a PK/PD model. | 6 hours
  The difference between observed and predicted values will be expressed as RMSE in percent.
Time required to achieve >30% decrease in PUAL compared to baseline. | 6 hours
  Time required for >30% decrease in PUAL will be expressed in minutes +/- standard deviation for each group.
To assess respiratory tolerance | 8 hours
  Using the respiratory rate and pulse oxygen saturation for respiratory tolerance
To assess neurological tolerance | 8 hours
  Using the Ramsay score for neurological tolerance
To assess hemodynamic tolerance | 8 hours
  Using the heart rate and blood pressure for hemodynamic tolerance
Measurement of administration comfort score using a visual analog scale ranging from 0 (maximum discomfort) to 10 (optimal comfort) (unitless). | 6 hours
  Administration comfort score will be expressed as mean +/- standard deviation for both groups.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Rouen, Rouen, France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barksdale AN, Hackman JL, Williams K, Gratton MC. ED triage pain protocol reduces time to receiving analgesics in patients with painful conditions. Am J Emerg Med. 2016 Dec;34(12):2362-2366. doi: 10.1016/j.ajem.2016.08.051. Epub 2016 Aug 27. PMID 27663766
- [Background] Gueant S, Taleb A, Borel-Kuhner J, Cauterman M, Raphael M, Nathan G, Ricard-Hibon A. Quality of pain management in the emergency department: results of a multicentre prospective study. Eur J Anaesthesiol. 2011 Feb;28(2):97-105. doi: 10.1097/EJA.0b013e3283418fb0. PMID 21119516
- [Background] Lvovschi V, Aubrun F, Bonnet P, Bouchara A, Bendahou M, Humbert B, Hausfater P, Riou B. Intravenous morphine titration to treat severe pain in the ED. Am J Emerg Med. 2008 Jul;26(6):676-82. doi: 10.1016/j.ajem.2007.10.025. PMID 18606320
- [Background] Galinski M, Robledo JB, Tellier E, Catoire P, De La Riviere C, Lvovschi V, Gil-Jardine C. Are Patients with Chronic Pain Less Satisfied with Their ED Management Than Non-Chronic Pain Patients? Am J Emerg Med. 2022 Jun;56:7-9. doi: 10.1016/j.ajem.2022.03.032. Epub 2022 Mar 19. No abstract available. PMID 35338897
- [Background] Mudd S. Intranasal fentanyl for pain management in children: a systematic review of the literature. J Pediatr Health Care. 2011 Sep-Oct;25(5):316-22. doi: 10.1016/j.pedhc.2010.04.011. Epub 2010 Jun 17. PMID 21867860
- [Background] Adelgais KM, Brent A, Wathen J, Tong S, Massanari D, Deakyne S, Sills MR. Intranasal Fentanyl and Quality of Pediatric Acute Care. J Emerg Med. 2017 Nov;53(5):607-615.e2. doi: 10.1016/j.jemermed.2017.05.027. Epub 2017 Sep 28. PMID 28967529
- [Background] Hudson RJ, Thomson IR, Henderson BT, Singh K, Harding G, Peterson DJ. Validation of fentanyl pharmacokinetics in patients undergoing coronary artery bypass grafting. Can J Anaesth. 2002 Apr;49(4):388-92. doi: 10.1007/BF03017328. PMID 11927479
- [Derived] Follet C, Dumont A, Roussel M, Gillibert A, Boedard C, Quillard M, Ruault S, Vallin F, Donnadieu N, Nunes Ferreira D, Pereira T, Joly LM, Lvovschi V, Duflot T. AEROfen: protocol for a phase I, open-label, randomised crossover study evaluating the efficiency of nebulised fentanyl in healthy volunteers - comparing facial versus intranasal administration via pharmacometric modelling. BMJ Open. 2025 Jul 3;15(7):e091125. doi: 10.1136/bmjopen-2024-091125. PMID 40615143